CLINICAL TRIAL: NCT03456466
Title: A Multi-center, Randomized, Double-blind, Parallel Control Clinical Trial to Assess the Similarity of the Safety and Pharmacokinetics of TQB2303 in Combination With Rituximab to Patients With AggressiveCD20 Positive Non-Hodgkin's Lymphoma
Brief Title: Study of TQB2303 in Patients With Aggressive CD20 Positive Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQB2303-I-01
Record Dates: First submitted 2017-12-23; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Non-hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: TQB2303 and Rituximab
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2303 (Experimental)
  Interventions: Drug: TQB2303
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: TQB2303 — 375mg/m2 ，iv
  Arms: TQB2303
Drug: Rituximab — 375mg/m2 ，iv
  Arms: Rituximab

SUMMARY:
Primary Outcome Measures:

Area under the curve (AUC) forTQB2303 and rituximab concentrations [ Time Frame: 85 days ]

Secondary Outcome Measures:

The Maximum Concentration (Cmax) of the TQB2303 and rituximab [ Time Frame: 85 days ] The area under the plasma concentration-time curve from 0 to inf (infinite) time (AUC0-∞); The time to reach the maximum plasma concentration after treatment (Tmax) Total clearance (CL); Elimination of half-life (t1 / 2); Apparent distribution volume (Vd).

ELIGIBILITY:
Inclusion Criteria:

1. Patients should participate in the study voluntarily and sign informed consent;
2. CD20-positive non-Hodgkin's lymphoma (NHL)：Diffuse Large B-cell Lymphoma；Mantle Cell Lymphoma；Follicular Lymphoma；Marginal Zone Lymphoma;
3. having obtained CR (complete remission) or CRu (uncertain complete remisson) after the prior therapy;And the investigators believe that CD20-positive B-cell NHL patients can benefit from anti-CD20 monoclonal antibody therapy;
4. aged from 18 to 75 years;
5. ECOG PS:0-1；
6. Life expectancy of more than 3 months

Exclusion Criteria:

1. Had received rituximab or other anti-CD20(+) monoclonal antibody treatment within 1 year before enrollment;
2. patients who were treated with antitumor therapy (including corticosteroid therapy) within 4 weeks prior to enrollment, or who had not recovered from the toxicity of the previous treatment;
3. Patients who participated in other clinical studies within 30 days ;
4. Serious hematologic dysfunction (white blood cell count of <3.0×10^9/L; absolute neutrophil count of <1.5×10^9/L; platelet count of < 75×10^9/L; hemoglobin level of <80g/L); In the absence of anticoagulant therapy, International Standardization Ratio (INR)> 1.5× ULN;Partial prothrombin time (PTT)Or activated partial thromboplastin time (aPTT)> 1.5 × ULN;) Hepatic dysfunction (total bilirubin level of > 1.5 × upper limit of normal (ULN); aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of > 2.0 × ULN;) renal dysfunction (serum creatinine level of > 1.5×ULN );
5. Other invasive malignancies except for cured the IB or lower level of cervical cancer; Non-invasive basal cells or squamous cell skin cancer; Get CR> 10 years of breast cancer;Get CR> 10 years of malignant melanoma;or other malignancies with CR> 5 years;
6. Central nervous system (CNS) lymphoma, AIDS-associated lymphoma;
7. Active infections and other serious non-malignant tumor diseases, Such as Qualitative pneumonia, Severe organic cardiovascular disease, Heart conduction block > 2,Myocardial infarction in 6 months, Cerebral infarction in 3 months,Cerebral hemorrhage,Thyroid dysfunction (TSH lower than the normal lower limit or higher than the upper limit of normal, and the researchers have a clinical significance);
8. Seropositive for HIV , HCV antibody; Or one of the following HBV findings :

   1. HBsAg positive;
   2. HBsAg negative, HBcAb positive and HBV DNA positive;
9. Plan major surgery, or surgical wound unhealed patients;
10. History of severe allergies, protein products and mouse products such as allergies;
11. Pregnancy or breast feeding. Companion for women of childbearing age or women of childbearing age,who reluctant to take appropriate contraceptive methods within one year after the last treatment of the study;Pregnancy before pregnancy screening, the women who blood / urine results were positive;
12. Receipt of a live/attenuated vaccine within 4 weeks prior to the Screening Visit;
13. Researchers think that do not fit into the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
AUC | 85 days
  Area under the curve (AUC) forTQB2303 and rituximab concentrations
Cmax | 85 days
  The Maximum Concentration (Cmax) of the TQB2303 and rituximab
AUC0-∞ | 85 days
  The area under the plasma concentration-time curve from 0 to inf (infinite) time
Tmax | 85 days
  The time to reach the maximum plasma concentration after treatment
CL | 85 days
  Total clearance
t1/2 | 85 days
  Elimination of half-life
Vd | 85 days
  Apparent distribution volume

SECONDARY OUTCOMES:
Evaluation of immunogenicity | 85 days
  Anti-drug antibody (ADA), neutralizing antibody (Nab detection when ADA positive)
Change of CD19+ CD20+ B-cells from baseline | 85 days
  Change of CD19+ CD20+ B-cells from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu